CLINICAL TRIAL: NCT02345473
Title: Detection and Clinical Significance of Circulating Cancer Cells in Patient Undergoing Radical Cystectomy
Acronym: CirCanCell
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Principal Investigator, Pagliarulo Vincenzo, Medical Doctor, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Other Study IDs: 4186
Record Dates: First submitted 2015-01-14; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Bladder Cancer; Circulating Tumor Cells
Keywords: Bladder cancer; Circulating cancer cells
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cystectomy patients: Arm of patients undergoing radical cystectomy for bladder cancer providing peripheral blood samples for detection of circulating cancer cells
  Interventions: Genetic: Detection of circulating tumor cells in blood samples
- Healthy volunteers: Arm of healthy subjects not undergoing radical cystectomy providing peripheral blood samples for detection of circulating cancer cells
  Interventions: Genetic: Detection of circulating tumor cells in blood samples

INTERVENTIONS:
Genetic: Detection of circulating tumor cells in blood samples — Ficoll based isolation of mononuclear cells from the peripheral blood of patients undergoing radical cystectomy, nucleic acids extraction and, finally, PCR based detection of sequences specific to cytokeratins.

SUMMARY:
Very few factors may be identified as prognostic for patients with bladder cancer undergoing radical cystectomy. Recently, detection of circulating tumor cells has shown to be very promising in anticipating both the likelyhood of distant metastases and survival in patients with breast cancer, melanoma, prostate cancer and other malignancies. In the present study we both tested the detection rate of circulating tumor cells using a PCR based methodology in the peripheral blood of patients undergoing radical cystectomy, and we further correlated our results with their clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Prior trans urethral resection of the bladder (TUR)
* Histological confirmation of a transitional cell carcinoma (TCC) of the bladder
* ECOG Performance Status ≤ 2
* WBC count ≥4,000/μL; platelet count ≥150,000/μL; creatinine ≤1.8 mg/dL; AST, ALT, and alkaline phosphatase ≤2X the upper limit of normal, normal total bilirubin
* recent (within 6 weeks of cystectomy) total body CT imaging study excluding distant metastases as well as upper urinary tract TCC

Exclusion Criteria:

* Neo-adjuvant chemotherapy (either planned or already performed)
* Patients receiving investigational medications
* Subjects not suitable for a radical cystectomy
* Patients not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing radical cystectomy for bladder cancer and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2005-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of circulating tumor cells | 8 years
  This outcome measure reflects the exact number of subjects diagnosed with circulating tumor cells within the total population of subjects included in the study

SECONDARY OUTCOMES:
Overall survival | 8 years
  Comparison of overall survival between the population of patients found with circulating tumor cells and those found without circulating tumor cells

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo VP Pagliarulo, Urologist, Principal Investigator — Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Locations (1):
- Vincenzo Pagliarulo, Bari, Italy, Italy

REFERENCES:
- [Background] Stein JP, Lieskovsky G, Cote R, Groshen S, Feng AC, Boyd S, Skinner E, Bochner B, Thangathurai D, Mikhail M, Raghavan D, Skinner DG. Radical cystectomy in the treatment of invasive bladder cancer: long-term results in 1,054 patients. J Clin Oncol. 2001 Feb 1;19(3):666-75. doi: 10.1200/JCO.2001.19.3.666. PMID 11157016
- [Background] Steven K, Poulsen AL. Radical cystectomy and extended pelvic lymphadenectomy: survival of patients with lymph node metastasis above the bifurcation of the common iliac vessels treated with surgery only. J Urol. 2007 Oct;178(4 Pt 1):1218-23; discussion 1223-4. doi: 10.1016/j.juro.2007.05.160. Epub 2007 Aug 14. PMID 17698113
- [Background] Madersbacher S, Hochreiter W, Burkhard F, Thalmann GN, Danuser H, Markwalder R, Studer UE. Radical cystectomy for bladder cancer today--a homogeneous series without neoadjuvant therapy. J Clin Oncol. 2003 Feb 15;21(4):690-6. doi: 10.1200/JCO.2003.05.101. PMID 12586807
- [Background] Lotan Y, Gupta A, Shariat SF, Palapattu GS, Vazina A, Karakiewicz PI, Bastian PJ, Rogers CG, Amiel G, Perotte P, Schoenberg MP, Lerner SP, Sagalowsky AI. Lymphovascular invasion is independently associated with overall survival, cause-specific survival, and local and distant recurrence in patients with negative lymph nodes at radical cystectomy. J Clin Oncol. 2005 Sep 20;23(27):6533-9. doi: 10.1200/JCO.2005.05.516. Epub 2005 Aug 22. PMID 16116151
- [Background] Attard G, Swennenhuis JF, Olmos D, Reid AH, Vickers E, A'Hern R, Levink R, Coumans F, Moreira J, Riisnaes R, Oommen NB, Hawche G, Jameson C, Thompson E, Sipkema R, Carden CP, Parker C, Dearnaley D, Kaye SB, Cooper CS, Molina A, Cox ME, Terstappen LW, de Bono JS. Characterization of ERG, AR and PTEN gene status in circulating tumor cells from patients with castration-resistant prostate cancer. Cancer Res. 2009 Apr 1;69(7):2912-8. doi: 10.1158/0008-5472.CAN-08-3667. PMID 19339269
- [Background] Marrinucci D, Bethel K, Bruce RH, Curry DN, Hsieh B, Humphrey M, Krivacic RT, Kroener J, Kroener L, Ladanyi A, Lazarus NH, Nieva J, Kuhn P. Case study of the morphologic variation of circulating tumor cells. Hum Pathol. 2007 Mar;38(3):514-9. doi: 10.1016/j.humpath.2006.08.027. Epub 2006 Dec 22. PMID 17188328
- [Background] Desgrandchamps F, Teren M, Dal Cortivo L, Marolleau JP, Bertheau P, Villette JM, Cortesse A, Teillac P, Le Duc A, Hamdy FC. The effects of transurethral resection and cystoprostatectomy on dissemination of epithelial cells in the circulation of patients with bladder cancer. Br J Cancer. 1999 Nov;81(5):832-4. doi: 10.1038/sj.bjc.6690771. PMID 10555753
- [Background] Osman I, Kang M, Lee A, Deng FM, Polsky D, Mikhail M, Chang C, David DA, Mitra N, Wu XR, Sun TT, Bajorin DF. Detection of circulating cancer cells expressing uroplakins and epidermal growth factor receptor in bladder cancer patients. Int J Cancer. 2004 Oct 10;111(6):934-9. doi: 10.1002/ijc.20366. PMID 15300806
- [Background] Ribal MJ, Mengual L, Marin M, Algaba F, Ars E, Fernandez PL, Oliva R, Villavicencio H, Alcaraz A. Molecular staging of bladder cancer with RT-PCR assay for CK20 in peripheral blood, bone marrow and lymph nodes: comparison with standard histological staging. Anticancer Res. 2006 Jan-Feb;26(1A):411-9. PMID 16475726
- [Background] Jiang J, Ulbright TM, Younger C, Sanchez K, Bostwick DG, Koch MO, Eble JN, Cheng L. Cytokeratin 7 and cytokeratin 20 in primary urinary bladder carcinoma and matched lymph node metastasis. Arch Pathol Lab Med. 2001 Jul;125(7):921-3. doi: 10.5858/2001-125-0921-CACIPU. PMID 11419977
- [Background] Chu P, Wu E, Weiss LM. Cytokeratin 7 and cytokeratin 20 expression in epithelial neoplasms: a survey of 435 cases. Mod Pathol. 2000 Sep;13(9):962-72. doi: 10.1038/modpathol.3880175. PMID 11007036
- [Background] Wu XR, Lin JH, Walz T, Haner M, Yu J, Aebi U, Sun TT. Mammalian uroplakins. A group of highly conserved urothelial differentiation-related membrane proteins. J Biol Chem. 1994 May 6;269(18):13716-24. PMID 8175808
- [Background] Wu X, Kakehi Y, Zeng Y, Taoka R, Tsunemori H, Inui M. Uroplakin II as a promising marker for molecular diagnosis of nodal metastases from bladder cancer: comparison with cytokeratin 20. J Urol. 2005 Dec;174(6):2138-42, discussion 2142-3. doi: 10.1097/01.ju.0000181214.32390.75. PMID 16280744
- [Background] Sawabata N, Okumura M, Utsumi T, Inoue M, Shiono H, Minami M, Nishida T, Sawa Y. Circulating tumor cells in peripheral blood caused by surgical manipulation of non-small-cell lung cancer: pilot study using an immunocytology method. Gen Thorac Cardiovasc Surg. 2007 May;55(5):189-92. doi: 10.1007/s11748-007-0101-2. PMID 17554991